CLINICAL TRIAL: NCT05237570
Title: Minimally Invasive Microsurgical Sinus-lift Through the Interradicular Septum. A Clinical Trial
Brief Title: Minimally Invasive Sinus Lift Through the Interradicular Septum
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2939/2020
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Bone Loss; Bone Loss, Age-related; Atrophy; Alveolar Process; Surgical Procedure, Unspecified
Keywords: maxillary sinus; sinus lift; xenograft
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): After the molar extraction, no intervention will be performed.
- Interradicular septum window group (Experimental): After the extraction of the molar, the maxillary sinus membrane will be elevated through a micro-window, previously done in the interradicular septum.
  Interventions: Procedure: Interradicular septum window

INTERVENTIONS:
Procedure: Interradicular septum window — In this group, the maxillary sinus will be accessed through a window in the interradicular septum and the membrane will be elevated, carrying out the regeneration of the area to facilitate subsequent implant placement.
  Arms: Interradicular septum window group

SUMMARY:
This study aims to describe a new approach for the reconstruction of the alveolar process in the sinus area. This minimally invasive approach will access the maxillary sinus through the alveolar process, elevating the sinus membrane in the area immediately above it. The regeneration may be achieved in the specific area required for dental implant placement, reducing the morbidity of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Plaque index and bleeding index less than 30%.
* Invagination of the sinus cavity in the interradicular area of the upper first molar.
* Upper first molar not restorable and with height of the interradicular remnant less than 5 mm.

Exclusion Criteria:

* Presence of systemic disease contraindicating the intervention.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-09-02 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Bone height | 9 months
  Bone height change

SECONDARY OUTCOMES:
Bucco-palatal bone width | 9 months
  Bucco-palatal bone width change

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moreno Rodriguez JA, Pecci-Lloret M, Ortiz Ruiz E, Ortiz Ruiz AJ. Preliminary Results of a Minimally Invasive Microsurgical Approach to Sinus Floor Elevation and Bone Reconstruction Using a Palatal Septum Window. Int J Periodontics Restorative Dent. 2021 Nov-Dec;41(6):e255-e263. doi: 10.11607/prd.4810. PMID 34818393